CLINICAL TRIAL: NCT05127226
Title: HALOS: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ION582 in Patients With Angelman Syndrome
Brief Title: HALOS: A Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Multiple Ascending Doses of ION582 in Participants With Angelman Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ION582-CS1; 2021-003009-23 (EudraCT Number)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1 MAD: Cohort A (Experimental): ION582 will be administered as IT injection over a period of 13 weeks, with a minimum of approximately 4 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 1 MAD: Cohort B (Experimental): ION582 will be administered as IT injection over a period of 13 weeks, with a minimum of approximately 4 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 1 MAD: Cohort C (Experimental): ION582 will be administered as IT injection over a period of 13 weeks, with a minimum of approximately 4 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 1 MAD: Cohort D (Experimental): ION582 will be administered as IT injection over a period of 13 weeks, with a minimum of approximately 4 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 1 MAD: Cohort E (Experimental): ION582 will be administered as IT injection of over a period of 13 weeks, with a minimum of approximately 4 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 1 MAD: Cohort F (Experimental): ION582 will be administered as IT injection over a period of 13 weeks, with a minimum of approximately 12 weeks between each dose administration.
  Interventions: Drug: ION582
- Part 2 Group 1 (Experimental): ION582 will be administered as IT injection of over a period of 49 weeks, with additional dosing intervals.
  Interventions: Drug: ION582
- Part 2 Group 2 (Experimental): ION582 will be administered as IT injection of over a period of 49 weeks, with additional dosing intervals.
  Interventions: Drug: ION582
- Part 3 Group 1 (Experimental): ION582 will be administered as IT injection of over a period of 145 weeks, with additional dosing intervals.
  Interventions: Drug: ION582
- Part 3 Group 2 (Experimental): ION582 will be administered as IT injection of over a period of 145 weeks, with additional dosing intervals.
  Interventions: Drug: ION582

INTERVENTIONS:
Drug: ION582 — ION582 will be administered by IT injection.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ascending doses of ION582 administered intrathecally in participants with Angelman syndrome.

DETAILED DESCRIPTION:
This is a Phase 1-2a, open-label study consisting of 3 parts in approximately 70 participants. Part 1 is a multiple ascending dose (MAD) study, consisting of a 13-week MAD Treatment Period and a minimum 12-week Post-MAD Follow-Up Period. Part 2 is a multi-center 49-week study where participants who completed Part 1 will receive IT bolus doses of ION582 followed by a minimum 12-week Part 2 follow up period. Part 3 extends the treatment period for participants who completed Part 2 for up to an additional 3 years followed by a 32-week post-LTE follow up period.

The study was amended in late 2025 to include a cohort of people with Angelman Syndrome under the age of 2 years old. Recruitment sites listed as "Recruiting" below are eligible to recruit individuals into this new cohort only. This page will continue to be updated to reflect the recruitment status of sites and the study. For more information, speak with your doctor or see the Study Contact information below.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant has a documented and certified diagnosis of Angelman syndrome (AS) (ubiquitin-protein ligase E3A [UBE3A] deletion or UBE3A mutation)
2. Male or female between the ages of 0-50 years of age, with signed informed consent from parent(s) or legal guardian(s)
3. Currently receiving stable standard of care treatments such as, stable doses of anti-epileptic medication, behavioral management medications, sleep medications, gabapentin, cannabidiol, and including special diets, supplements or nutritional support for at least 3 months prior to first dose.
4. Follow good study practice and not participate in the sharing of personal or study information on social media platforms, such as any website or social media site (e.g., Facebook, Instagram, Twitter, YouTube, etc.) until notified that the study is completed.

Key Exclusion Criteria:

1. Has documented molecular AS confirmation of paternal uniparental disomy (UPD) or imprinting defect (ID).
2. Any clinically significant (CS) cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurologic, malignant, metabolic, psychiatric, or other condition that, in the judgment of the Investigator, will pose a safety risk, will make the patient unsuitable for participation in, and/or unable to complete the study procedures. Has poorly controlled seizures as determined by the Investigator or has documented Status Epilepticus in the past 6 months that could pose a safety risk while on study.
3. Known bone, spine, bleeding, or other disorder that exposes the patient to risk of injury or unsuccessful lumbar puncture. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid, antisense oligonucleotide [ASOs]). COVID-19 vaccinations are allowed.
4. Any prior use of gene therapy. Have any other conditions, which, in the opinion of the Investigator would make the participant unsuitable for inclusion or could interfere with the participant taking part in or completing the study.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple doses of ION582 (incidence, severity, and dose-relationship of adverse effects and changes in the laboratory parameters). | Part 1: Up to Week 45; Part 2: Up to Week 81
  The safety and tolerability of ION582 will be assessed by determining the incidence, severity, and dose relationship of adverse effects and changes in the laboratory parameters by dose.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ION582 | Part 1: Up to Week 45; Part 2: Up to Week 81
Time to Reach Maximal Plasma Concentration (Tmax) of ION582 | Part 1: Up to Week 45; Part 2: Up to Week 81
Plasma Elimination Half-Life (t1/2λz) of ION582 | Part 1: Up to Week 45; Part 2: Up to Week 81
Concentration ION582 in CSF | Part 1: Up to Week 13; Part 2: Up to Week 49

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - Rady Children's Hospital, San Diego, California
  - Colorado Children's Hospital Research Institute, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill School of Medicine, Carrboro, North Carolina
  - Texas Children's Hospital, Houston, Texas
- Sydney Children's Hospital, Kids Cancer Centre, Randwick, Australia
- Necker-Enfants Malades Hospital, Paris, France
- Sheba Medical Center, Ramat Gan, Israel
- Azienda Ospedaliera Universitaria Pisana, Pisa, Italy
- STRONG Group University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/